CLINICAL TRIAL: NCT00048009
Title: Evaluation of Various Doses of Ro 27-2771 (Test Drug) in Asthmatic Patients Not Treated With Inhaled Corticosteroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: BA16631
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Dual Integrin Antagonist

SUMMARY:
The purpose of this study is to determine the appropriate dose of Ro 27-2441 (test drug) to be used in future studies, assess the efficacy and safety, and the anti-inflammatory action of the test drug in the treatment of asthmatic patients who are not currently receiving chronic therapy with corticosteroids. The research is being conducted at up to 80 clinical research sites in the US, Mexico, and Canada. Study participants will have a number of visits to a research site over approximately a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma for more than one year
* Current treatment for asthma with short acting inhaled beta 2 agonists (such as albuterol) only
* In good health ad demonstrated by medical history and physical exam
* Negative urine pregnancy test
* Commitment to use two forms of effective contraception simultaneously throughout the study duration and for one month after discontinuing therapy

Exclusion Criteria:

* Asthma necessitating treatment with inhaled corticosteroids for at least one month before the start of the study
* History of severe asthma necessitating the use of oral/injectable corticosteroids within the last 2 months and/and or two bursts in the last year
* Undergoing allergy shots unless on a stable maintenance dose for three months before the start of the study
* History of chronic pulmonary diseases other than asthma
* Treatment of conditions other than asthma with oral corticosteroids within one month of the start of the study
* Current tobacco use
* Smoking history of greater than 10 pack-year history of cigarette smoking (number of packs smoked per day times the number of years smoked)
* History or evidence of drug or alcohol abuse
* Diagnosis or evidence of an infectious illness within one month of Visit 1
* Clinically significant diseases as assessed by the study doctor
* Participation in another clinical study with an experimental drug within one month of start of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10-25 (Actual); Primary Completion 2004-02-02 (Actual); Study Completion 2004-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (60):
  - Scottsdale, Arizona
  - Huntington Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Palmdale, California
  - San Diego, California
  - San Jose, California
  - Walnut Creek, California
  - Denver, Colorado
  - Louisville, Colorado
  - Wheat Ridge, Colorado
  - Hartford, Connecticut
  - Tallahassee, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Normal, Illinois
  - River Forest, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lenexa, Kansas
  - Metairie, Louisiana
  - North Dartmouth, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Cherry Hill, New Jersey
  - Princeton, New Jersey
  - Teaneck, New Jersey
  - Farmingdale, New York
  - Rochester, New York
  - Rockville Centre, New York
  - Elizabeth City, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Murray, Utah
  - Kirkland, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Wenatchee, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (6):
  - Adelaide
  - Brisbane
  - Melbourne
  - Perth
  - Sydney
  - Woodville
- Canada (5):
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Mexico (7):
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - Mérida
  - México
  - Monterrey
  - Puebla City
- Ponce, Puerto Rico